CLINICAL TRIAL: NCT07298889
Title: Effect of High Versus Low Positive End-Expiratory Pressure on Intubation-Free Survival in Patients With Pneumonia or ARDS Receiving Noninvasive Ventilation: A Multicenter Randomized Controlled Trial
Brief Title: High PEEP in Noninvasive Ventilation Patients With Pneumonia or ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, attending physician, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingMU06
Record Dates: First submitted 2025-12-08; First posted 2025-12-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Noninvasive Ventilation; Pneumonia; ARDS
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High PEEP group (Experimental): Patients in high PEEP group will received 10 to 15 cmH2O of PEEP during noninvasive ventilation.
  Interventions: Procedure: The level of PEEP during noninvasive ventilation
- Low PEEP group (Active Comparator): Patients in low PEEP group will received 5 cmH2O of PEEP during noninvasive ventilation.
  Interventions: Procedure: The level of PEEP during noninvasive ventilation

INTERVENTIONS:
Procedure: The level of PEEP during noninvasive ventilation — In patients receiving noninvasive ventilation, participants will be randomly assigned to either a low or a high PEEP group. In the high PEEP group, PEEP will be set between 10 and 15 cmH2O. In the low PEEP group, PEEP will be maintained at 5 cmH2O.

SUMMARY:
Noninvasive ventilation is commonly employed in patients with pneumonia or acute respiratory distress syndrome (ARDS) and has been shown to reduce the need for intubation and invasive mechanical ventilation. However, the rate of noninvasive ventilation failure remains substantial, at approximately 40%. Compared with patients in whom noninvasive ventilation succeeds, those who experience noninvasive ventilation failure have a higher likelihood of mortality during their intensive care unit or hospital stay. Therefore, improving the success rate of noninvasive ventilation is clinically important. In patients with lung consolidation receiving invasive mechanical ventilation, high positive end-expiratory pressure (PEEP) can improve oxygenation. Noninvasive ventilation operates on similar physiological principles and can also deliver high PEEP via a mask interface. Nevertheless, there is limited evidence regarding the use of high PEEP during mask-delivered noninvasive ventilation. This study aimed to evaluate whether high PEEP can increase intubation-free survival in patients with pneumonia or ARDS who are treated with noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* PaO2/FiO2 ≤300 mmHg or SpO2/FiO2 ≤315（SpO2 ≤97%)
* Anticipated NIV duration > 12 h
* Preserved consciousness (GCS≥13)

Exclusion Criteria:

* Use of NIV > 24 h before randomization
* Acute-on-chronic respiratory failure
* Congestive heart failure
* Use of NIV after extubation (within 48 hours)
* Contraindications to NIV (e.g., anatomical malformations, recent pulmonary/esophageal surgery [within 7 days])
* Pneumothorax
* NIV intolerance
* Refusal to participate
* Pregnancy
* Need for emergency intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2026-01-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day intubation-free survival | from randomization to 28 days after randomization

SECONDARY OUTCOMES:
28-day intubation rate | from randomization to 28 days after randomization
the need for intubation within 28 days | from randomization to 28 days after randomization
  The rate of the need for intubation within 28 days after randomization was assessed by two independent reviewers with extensive critical care experience.
28-day survival | from randomization to 28 days after randomization
7-category ordinal scale for clinical improvement at 28 days | from randomization to 28 days after randomization
  The 7-category ordinal scale is as follows: 1 = not hospitalized and has resumed normal activities; 2 = not hospitalized but unable to resume normal activities; 3 = hospitalized without requiring supplemental oxygen; 4 = hospitalized and requiring supplemental oxygen; 5 = hospitalized and requiring HFNC, NIV, or both; 6 = hospitalized and requiring extracorporeal membrane oxygenation (ECMO), invasive mechanical ventilation, or both; 7 = death.
28-day invasive ventilator-free days | from randomization to 28 days after randomization
28-day noninvasive ventilator days | from randomization to 28 days after randomization
Length of ICU stay | up to 24 weeks
Length of hospital stay | up to 24 weeks
ICU mortality | up to 24 weeks
Hospital mortality | up to 24 weeks
60-day mortality | from randomization to 60 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
These study data contain ethnic demographic information. Since it remains unclear whether Chinese laws permit the public disclosure of such data upon the completion of the research, a decision has been made to temporarily withhold data sharing during the study design phase.